CLINICAL TRIAL: NCT05364398
Title: Does Stump-Preserving Anterior Cruciate Ligament Reconstruction Provide Better Functional Outcomes?
Brief Title: Comparison of ACL Reconstruction With Stump Preservation and Stump Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed El-Desouky, Associate Professor of Orthopedic surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-09-2017
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Knee Ligament Injury
Keywords: Anterior cruciate ligament reconstruction; tibial stump; stump preservation; knee proprioception.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL reconstruction with stump preservation (Active Comparator)
  Interventions: Procedure: ACL reconstruction
- ACL reconstruction with stump resection (Active Comparator)
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — Use of hamstring tendons graft to replace the torn ACL and being passed and fixed through the femoral and tibial sides

SUMMARY:
To assess the clinical outcome in patients who had ACL reconstruction with preservation of the remnant and compare it with patients in whom the stump was resected

DETAILED DESCRIPTION:
100 patients are subjected to ACL reconstruction. Half of them had ACL reconstruction with Stump preservation and the other half had ACL reconstruction with stump resection.

The clinical outcome in both groups is assessed and compared

ELIGIBILITY:
Inclusion Criteria:

* patients with torn ACL within 6 months

Exclusion Criteria:

* Old ACL injury Multi-ligamentous knee injuries Mal-alignments

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Knee stability | 2 years
  KT-1000 Arthrometer
Knee proprioception | 2 years
  Passive angle reproduction test
Lysholm score | 2 years
Tegner activity score | 2 years
IKDC score | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Desouky MA, Ezzat M, Abdelrazek BH. Clinical outcomes in stump-preserving versus stump-sacrificing anterior cruciate ligament reconstruction; a randomized controlled study. BMC Musculoskelet Disord. 2022 Jul 23;23(1):703. doi: 10.1186/s12891-022-05665-3. PMID 35870924